CLINICAL TRIAL: NCT04012216
Title: Sleep Respiratory Disorders in Patients With Moderate to Severe Persistent Rhinitis: a Prospective, Predictive Study
Brief Title: Sleep Respiratory Disorders in Patients With Moderate to Severe Persistent Rhinitis
Acronym: JawRhin1
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: ADENE (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0473
Record Dates: First submitted 2019-06-27; First posted 2019-07-09 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population: Patients consulting for persistant, moderate-to-severe rhinitis and meeting eligibility criteria.
  Interventions: Device: Measure of mandibular movement using a mid-sagittal magnetic sensor (Brizzy, Jawac©) Nomics, Liege, Belgium); Device: Gold standard: polysomnography

INTERVENTIONS:
Device: Measure of mandibular movement using a mid-sagittal magnetic sensor (Brizzy, Jawac©) Nomics, Liege, Belgium) — A mid-sagittal MM magnetic sensor (Brizzy, Jawac©) Nomics, Liege, Belgium) measures the distance in mm between two parallel, coupled, resonant circuits placed on the forehead and on the chin. Measurements last one night.
Device: Gold standard: polysomnography — Polysomnography will be performed according to the American Academy of Sleep Medicine Recommendations 2018

SUMMARY:
The general aim of this study is to demonstrate that the measurement of respiratory effort assessed by mandibular movements during sleep is a useful measure for the screening of sleep disordered breathing (SDB) in patients with moderate to severe persistent rhinitis (R). The primary objective is therefore to determine a mandibular movement respiratory disturbance index (MM-RDI) threshold associated with a polysomnography respiratory disturbance index (PSG-RDI) ≥ 15 / h in a population of patients with moderate-to-severe persistent R.

DETAILED DESCRIPTION:
The secondary objectives of the study are to evaluate the concordance and correlation between:

* MM-RDI,
* the respiratory effort evaluated by MM,
* polysomnography (PSG) results,
* quality of life questionnaires,
* clinical data,
* treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient consulting for persistant, moderate-to-severe rhinitis
* The patient has signed the informed consent
* The patient is a beneficiary of a social security programme (national health insurance)
* Patient living in the Montpellier region (< 30 kilometers).

Exclusion Criteria:

* The patient is participating in another study that precludes participation in the present study
* The patient is in an exclusion period determined by another study
* It is impossible to correctly inform the patient
* The patient cannot fluently read French
* Vulnerable patient populations according to French Health Code article L1121-6
* Adult under guardianship or incapable of giving consent according to French Health Code article L1121-8
* Pregnancy, breastfeeding (French Health Code article L1121-5)
* Any element that renders participation in the study problematic according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting for persistant, moderate-to-severe rhinitis.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
The mandibular movement respiratory disturbance index | Day 7
The polysomnography respiratory disturbance index | Day 7

SECONDARY OUTCOMES:
Epworth scale score | Day 1
  This questionnaire describes sleepiness with a score that ranges from 0 to 24. Higher scores indicate more sleepiness.
Epworth scale score | Day 7
  This questionnaire describes sleepiness with a score that ranges from 0 to 24. Higher scores indicate more sleepiness.
The Karolinska questionnaire | Day 1
  The complete name of this questionnaire is the "Karolisnska questionnaire." This questionnaire describes sleepiness when the patient is driving. No total score reported. The minimum score is 1 and the maximal score is 9. The best outcome is 1 (patient is extremely vigilant), the worst outcome is 9 (very sleepy, takes great effort to stay awake, fights against sleep).
The Karolinska questionnaire | Day 7
  The complete name of this questionnaire is the "Karolisnska questionnaire." This questionnaire describes sleepiness when the patient is driving. No total score reported. The minimum score is 1 and the maximal score is 9. The best outcome is 1 (patient is extremely vigilant), the worst outcome is 9 (very sleepy, takes great effort to stay awake, fights against sleep).
The Pittsburgh Sleep Quality Index (PSQI) | Day 7
  The Pittsburg Sleep Quality Index (PSQI) measures the quality of sleep. It contains 19 self-rated questions and 5 questions by the bed partner or roommate (if one is available). Only self -rated questions are included in the scoring. The 19 self-rated items are combined in seven component scores each of which has a range of 0-3 points. In all the cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas. The 7 components are subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication and daytime dysfunction.
The mobility dimension of the EQ-5D-3L Questionaire (the 3-level version of Euroqol EQ-5D) | Day 1
  The Euro Quality Of Life-5 dimensions - 3 levels (EQ-5D-3L) scale is a descriptive system comprising the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. In addition, there is a visual analogue scale (VAS) to indicate the general health status with "0" indicating the worse health and "100" indicating the best health.
The autonomy dimension of the EQ-5D-3L Questionaire (the 3-level version of Euroqol EQ-5D) | Day 1
  The Euro Quality Of Life-5 dimensions - 3 levels (EQ-5D-3L) scale is a descriptive system comprising the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. In addition, there is a visual analogue scale (VAS) to indicate the general health status with "0" indicating the worse health and "100" indicating the best health.
The daily activities dimension of the EQ-5D-3L Questionaire (the 3-level version of Euroqol EQ-5D) | Day 1
  The Euro Quality Of Life-5 dimensions - 3 levels (EQ-5D-3L) scale is a descriptive system comprising the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. In addition, there is a visual analogue scale (VAS) to indicate the general health status with "0" indicating the worse health and "100" indicating the best health.
The pain dimension of the EQ-5D-3L Questionaire (the 3-level version of Euroqol EQ-5D) | Day 1
  The Euro Quality Of Life-5 dimensions - 3 levels (EQ-5D-3L) scale is a descriptive system comprising the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. In addition, there is a visual analogue scale (VAS) to indicate the general health status with "0" indicating the worse health and "100" indicating the best health.
The anxiety-depression dimension of the EQ-5D-3L Questionaire (the 3-level version of Euroqol EQ-5D) | Day 1
  The Euro Quality Of Life-5 dimensions - 3 levels (EQ-5D-3L) scale is a descriptive system comprising the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. In addition, there is a visual analogue scale (VAS) to indicate the general health status with "0" indicating the worse health and "100" indicating the best health.
The visual analog scale from the EQ-5D-3L Questionaire (the 3-level version of Euroqol EQ-5D) | Day 1
  The Euro Quality Of Life-5 dimensions - 3 levels (EQ-5D-3L) scale is a descriptive system comprising the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. In addition, there is a visual analogue scale (VAS) to indicate the general health status with "0" indicating the worse health and "100" indicating the best health.
  "0" score is the minimum value, "100" score is the maximum value. There is no subscale. The better outcome is "100" (100 indicating the best health status)
The Nasal Obstruction Symptom Evaluation (NOSE) questionnaire | Day 1
  The NOSE questionnaire is composed of five subscales, namely: 1) nasal congestion or stuffiness; 2) nasal blockage or obstruction; 3) trouble breathing through my nose; 4) trouble sleeping; 5) unable to get enough air through my nose during exercise or exertion.
  All subscales are scored using a 5-point Likert scale ranging from 0 to 4 (0=not a problem, 1=very mild problem, 2=moderate problem, 3=fairly bad problem, 4=severe problem). Each definitive subscale score is obtained after multiplying the Likert score by five. All subscales are added to give a total score (total score range from 0 (no nasal obstruction) to 100 (the most severe nasal obstruction).
The Nasal Obstruction Symptom Evaluation (NOSE) questionnaire | Day 7
  The NOSE questionnaire is composed of five subscales, namely: 1) nasal congestion or stuffiness; 2) nasal blockage or obstruction; 3) trouble breathing through my nose; 4) trouble sleeping; 5) unable to get enough air through my nose during exercise or exertion.
  All subscales are scored using a 5-point Likert scale ranging from 0 to 4 (0=not a problem, 1=very mild problem, 2=moderate problem, 3=fairly bad problem, 4=severe problem). Each definitive subscale score is obtained after multiplying the Likert score by five. All subscales are added to give a total score (total score range from 0 (no nasal obstruction) to 100 (the most severe nasal obstruction).
The Allergic Rhinitis Control Test (ARCT) rhinitis questionnaire | Day 1
  The Allergic Rhinitis Control Test (ARCT is a self-completion questionnaire assessing the control of chronic rhinitis. It is made up of five questions scored from 1 to 5, and these individual scores are then added up to obtain a score ranging from 5 (worse score) to 25 (best score). The five questions are: during the last 2 weeks, has your allergic rhinitis had an effect on your professional/personal activities ; during the last 2 weeks, has your allergic rhinitis made you irritable ; during the last 2 weeks, has your allergic rhinitis disturbed your sleep (going to sleep, waking at night) ; during the last 2 weeks, have you needed to use an additional treatment not prescribed by your doctor to treat your allergic rhinitis ; during the last 2 weeks, how would you assess your allergic rhinitis.
Total sleep time (TST) | Day 7
  From polysomnography.
Obstructive apnea index | Day 7
  From polysomnography.
Mixed apnea index | Day 7
  From polysomnography.
Apnea index | Day 7
  From polysomnography.
Hypopnea index | Day 7
  From polysomnography.
Apnea and Hypopnea index | Day 7
  From polysomnography.
Respiratory effort related arousal index | Day 7
  From polysomnography.
Respiratory Disturbance Index | Day 7
  From polysomnography.
Time spent snoring | Day 7
  From polysomnography.
Oxygen desaturation ≥ 3% index | Day 7
  From polysomnography.
Time below 90% SpO2 | Day 7
  From polysomnography.
% of TST below 90% of SpO2 | Day 7
  From polysomnography.
Mean SpO2 | Day 7
  From polysomnography.
Minimal SpO2 during sleep | Day 7
  From polysomnography.
Time in bed | Day 7
  From polysomnography.
Sleep Onset Latency | Day 7
  From polysomnography.
Wake After Sleep Onset (WASO) | Day 7
  From polysomnography.
Wake During Sleep Period | Day 7
  From polysomnography.
Sleep Latency | Day 7
  From polysomnography.
Random eye movement (REM) stage latency | Day 7
  From polysomnography.
Percentage of sleep efficiency | Day 7
  From polysomnography.
Time in sleep stage | Day 7
  From polysomnography.
Percent of TST in sleep stage | Day 7
  From polysomnography.
Arousal index | Day 7
  From polysomnography.
Arousal index associated with respiratory events | Day 7
  From polysomnography.
The periodic limb movement (PLM) index | Day 7
  From polysomnography.
PLM arousal | Day 7
  From polysomnography.
Number of limb movements associated with respiratory events index | Day 7
  From polysomnography.
Photoplethysmography arousal index | Day 7
  From polysomnography.
Signal validity | Day 7
  From mandibular movement recordings.
TST | Day 7
  From mandibular movement recordings.
WASO | Day 7
  From mandibular movement recordings.
% of TST spent in respiratory effort | Day 7
  From mandibular movement recordings.
Respiratory fragmentation of sleep index | Day 7
  From mandibular movement recordings.
Fragmentation of sleep index | Day 7
  From mandibular movement recordings.
ARIA rhinitis classification | Day 1
  ARIA = Allergic Rhinitis and its Impact on Asthma
Presence/absence of asthma | Day 1
  Does the patient have asthma? yes/no
For asthma patients, the GINA control score | Day 1
  GINA = Global Initiative for Asthma
Forced expiratory volume in 1 second, % predicted | Day 1
  From spirometry.
Forced vital capacity, % predicted | Day 1
  From spirometry.
Forced expiratory volume in 1 second / Forced vital capacity (% litres/litres)predicted | Day 1
  From spirometry.
Forced expiratory volume 25-75, % predicted predicted | Day 1
  From spirometry.
Antecedent of public road or work accident (yes/no) | Day 1
Patient reports presence/absence of poor sleep | Day 1
Patient reports presence/absence of snoring | Day 1
Patient reports presence/absence of dry mouth | Day 1
Patient reports presence/absence of concentration difficulty | Day 1
Patient reports presence/absence of headaches | Day 1
Allergen prick test results | Day 1
List of concomitant medications | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Dany JAFFUEL, MD, PhD, Principal Investigator — Department of Respiratory Medicine and Addiction Medicine
Locations (1):
- Chu Montpellier, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to make the study data available to interested researchers as well as to provide proof of transparency for the study. Data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
  Data will be made available to the public on a not-for-profit, free platform that allows access control (zenodo.org). Links on osf.io/clinicaltrials.gov will point towards the upload.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As close to "real time" as possible, the following supporting information will be made public:
  * Study Protocol
  * Statistical Analysis Plan
  * Participant Information Materials
  * Clinical Study Report
  * Analytic code
  These will be posted and registered on osf.io/clinicaltrials.gov.
  Individual datasets will be made available to reviewers at time of submission. Full public access to data will be implemented within 4 weeks following publication acceptation.
Access Criteria: The conditions under which members of the public will be granted access (via zenodo.org) to the uploaded files are:
  * The data will be used/examined in a not-for-profit manner;
  * The data will not be used in an attempt to identify a participant or group of participants;
  * The user does not work for a private insurance company;
  * The data will not be used in support of any kind of private insurance policy or health penalties;
  * The data will be used/examined for the advancement of science/teaching while respecting participant/patient privacy and rights;
  * The user will state why they wish to access the data.
URL: https://osf.io/whfdc/